CLINICAL TRIAL: NCT07399548
Title: Effects of Plyometric Training on Linear Sprint, Change-of-Direction, and Isokinetic Strength Performances in Male Basketball Players
Brief Title: Effects of 8-Week Plyometric Training on Basketball Performance and Isokinetic Strength
Acronym: PT-BASKET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Mustafa Şakir Akgül, Department Head of Sports Management, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-2287; 2025-2287 (Other: Kastamonu University)
Record Dates: First submitted 2026-02-01; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Athletic Performance; Physical Fitness; Muscle Strength; Plyometric Exercise Adaptations; Neuromuscular Performance in Athletes
Keywords: Plyometric Training; Basketball Performance; Change of Direction; Linear Sprint Velocity
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: The study followed a pre-test/post-test parallel-group randomized design. A total of 24 male basketball players were assigned to one of two arms: 1. Experimental Group (n = 12): Participants integrated a progressive plyometric training (PT) program into their routine basketball schedule. The PT was performed twice weekly (Tuesdays and Thursdays) for 8 weeks, focusing on high-intensity jumping and bounding exercises to enhance the stretch-shortening cycle. 2. Control Group (n = 12): Participants continued their standard basketball training program (technical and tactical drills) without any additional plyometric intervention. Both groups were assessed simultaneously at baseline (Week 0) and post-intervention (Week 8) using the same testing battery (25-meter sprint, V-cut agility, countermovement jump, and isokinetic dynamometry) under identical environmental conditions to ensure comparability.
Masking Description: Due to the nature of the intervention (physical exercise and plyometric training), it was not possible to mask the participants or the coaching staff to the group assignments. Both the experimental and control groups were aware of their respective training protocols. However, to minimize bias during the assessment and data processing phases: 1.Data Analysis: The statistical analysis was performed by a researcher who was blinded to the group allocations. All data were coded to ensure anonymity until the completion of the analysis. 2. Standardization: To ensure objectivity, all physical performance tests, including the 25-meter sprint, V-cut agility, and isokinetic strength, were conducted using automated electronic timing systems (Witty, Microgate, Italy) and computerized dynamometers (Isomed 2000, D&R Ferstl GmbH, Germany). These objective measures eliminate potential manual measurement errors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental): Participants in the Experimental Group (EG) followed a structured, progressive 8-week plyometric training (PT) program integrated into their regular basketball routine. The intervention was administered twice weekly (Tuesdays and Thursdays) with at least 48 hours of recovery between sessions. The program included vertical, horizontal, and lateral movements such as countermovement jumps (CMJ), box jumps, depth jumps, lateral bounds, and squat jumps. The volume progressed from 80 ground contacts per session in the first two weeks to 140 ground contacts per session in the final two weeks. Exercises were performed at maximal effort to maximize the utilization of the stretch-shortening cycle (SSC). All sessions were supervised by a certified strength and conditioning specialist to ensure proper technique and safety. This program was performed in addition to their standard technical and tactical basketball drills, which were identical to those performed by the control group.
  Interventions: Other: 8-Week Progressive Plyometric Training Program
- Standard Basketball Training (No Intervention): Participants in the Control Group (CG) followed their standard basketball training routine for a duration of 8 weeks. This arm serves as the baseline to compare the specific effects of the plyometric intervention administered to the experimental group. The sessions consisted of standard technical and tactical basketball drills, including shooting practice, defensive positioning, offensive sets, and scrimmages (e.g., 3-on-3 or 5-on-5 games). Participants maintained their regular schedule of five training sessions per week, with each session lasting approximately 90 to 120 minutes. Participants in this group did not participate in any structured plyometric, strength, or power-based conditioning programs during the study period. All participants were instructed to maintain their normal nutritional habits and daily physical activities to ensure that no external variables influenced the performance outcomes.

INTERVENTIONS:
Other: 8-Week Progressive Plyometric Training Program — The intervention consists of a structured 8-week progressive plyometric training (PT) program designed specifically for competitive basketball players. It is performed twice weekly as a supplement to standard technical and tactical basketball drills.
  1. Progressive Volume: The training dosage is strictly controlled based on ground contacts per session, progressing from 80 contacts during Weeks 1 to 2, up to 140 contacts during Weeks 7 to 8.
  2. Movement Protocols: The protocol includes multi-planar movements such as vertical (box jumps, countermovement jumps), horizontal (broad jumps), and lateral (lateral bounds) exercises to simulate basketball-specific demands.
  3. Execution & Recovery: Exercises are performed at maximal effort, focusing on minimizing ground contact time to optimize the stretch-shortening cycle (SSC). Sessions occur on a standard basketball court for surface adaptation. A recovery period of 48 to 72 hours is provided between sessions to prevent overtraining.
  Other Names: Plyometric Training; Stretch-Shortening Cycle Training; Lower-Body Power Training; Explosive Strength Training
  Arms: Plyometric Training

SUMMARY:
This study aims to evaluate the effects of an 8-week plyometric training program on the physical performance of male basketball players. The research focuses on measuring improvements in linear sprinting speed, change-of-direction (agility) abilities, and vertical jump height. Additionally, the study examines changes in the participants' muscle strength through isokinetic testing. Twenty-four trained basketball players were divided into two groups: the control group followed their regular basketball training, while the experimental group added specific plyometric exercises, such as jumps and bounds, twice per week. By comparing the results before and after the 8-week intervention period, the study seeks to determine if this training method effectively enhances the athletic skills required in competitive basketball.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to investigate the multidimensional effects of a structured plyometric training (PT) intervention on competitive male basketball players. While vertical jump performance is a common focus in PT research, this study specifically evaluates the transfer of adaptations to sport-specific locomotor tasks and isokinetic muscle strength profiles.Participants (N = 24) were randomly assigned to either an experimental group (EG) or a control group (CG). Both groups maintained their standard basketball training, including shooting, 3-on-3 games, and defensive drills. The EG performed an additional 8-week progressive plyometric program twice weekly, consisting of exercises such as box jumps, depth jumps, and bounding, with a total volume ranging from 80 to 140 ground contacts per session. Training volume was meticulously logged, and an adherence rate of at least 85% was required for inclusion in the final analysis.Performance was evaluated through a comprehensive testing battery conducted pre- and post-intervention under standardized conditions. The primary outcomes focused on linear sprint speed (25-meter sprint) and change-of-direction (CoD) ability (V-cut test), which are critical for the high-intensity demands of basketball. Secondary outcomes included vertical jump height measured via countermovement jump (CMJ) with and without arm swing, and isokinetic knee and hip strength assessed at angular velocities of 60 degrees per second and 180 degrees per second.The study hypothesized that the addition of PT would lead to superior gains in sprint and CoD performance compared to basketball training alone. Furthermore, it aimed to explore whether these performance improvements are accompanied by significant changes in isokinetic torque production. Data were analyzed using a 2 (Time) x 2 (Group) repeated-measures ANOVA to identify significant interactions. Normality was verified using Skewness and Kurtosis z-scores, with Winsorization applied to outliers to maintain data robustness.

ELIGIBILITY:
Inclusion Criteria:

* Active and licensed male basketball players.
* Age between 18 and 22 years.
* Minimum of 3 years of competitive basketball experience.
* Currently participating in regular team training at least 5 days per week.
* Free from any lower-limb musculoskeletal injuries for at least 6 months prior to the study.

Exclusion Criteria:

* Presence of any acute or chronic injury that limits maximal performance during the study period.
* Concurrent participation in any other external strength or power training programs.
* Failure to attend more than 10 percent of the intervention sessions.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
25-meter Linear Sprint Time | Baseline (Week 0) and Post-intervention (Week 8).
  Time taken to complete a 25-meter straight-line sprint from a standing start. This measure evaluates linear speed and explosive acceleration. The test is conducted on a basketball court using electronic timing gates, with the best time of three trials recorded to ensure data accuracy.
V-cut Agility Test Time | Baseline (Week 0) and Post-intervention (Week 8).
  Time taken to complete the V-cut agility test, which requires participants to perform four 25-degree directional changes over a 20-meter distance. This measure evaluates change-of-direction speed and maneuverability. The best time of three trials is recorded in seconds using electronic timing gates.

SECONDARY OUTCOMES:
Countermovement Jump (CMJ) Height | Baseline (Week 0) and Post-intervention (Week 8).
  Assessment of explosive lower-body power. Measured using an Optojump photoelectric system (Microgate, Italy) while participants perform a maximal vertical jump with hands on hips.
Isokinetic Peak Torque of Knee Extensors and Flexors | Baseline (Week 0) and Post-intervention (Week 8).
  Maximal concentric muscle strength of the knee extensors and flexors is measured at angular velocities of 60 degrees per second and 180 degrees per second. Assessments are performed using an isokinetic dynamometer (Isomed 2000, D&R Ferstl GmbH, Germany). The peak torque value from five maximal repetitions at each speed is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Faculty of Sports Sciences, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant dataset, including performance outcomes (25m sprint, V-cut agility, vertical jump, and isokinetic strength values), will be made available to researchers upon reasonable request. Interested parties must provide a methodologically sound research proposal and sign a data access agreement. Requests should be directed to the Principal Investigator at Kastamonu University
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available starting 6 months after article publication and will remain accessible for up to 36 months.
Access Criteria: Data will be shared with investigators who provide a methodologically sound proposal to achieve the aims in the approved proposal. Requests should be directed to the corresponding author.

REFERENCES:
- [Result] Ramirez-Campillo R, Perez-Castilla A, Thapa RK, Afonso J, Clemente FM, Colado JC, de Villarreal ES, Chaabene H. Effects of Plyometric Jump Training on Measures of Physical Fitness and Sport-Specific Performance of Water Sports Athletes: A Systematic Review with Meta-analysis. Sports Med Open. 2022 Aug 29;8(1):108. doi: 10.1186/s40798-022-00502-2. PMID 36036301
- See also: Institutional website of the Faculty of Sports Sciences where the study was conducted. — https://sporbilimleri.kastamonu.edu.tr/